CLINICAL TRIAL: NCT04766983
Title: Cohort Study to Evaluate the Incidence of Ventilator-associated Pneumonia by Means of Bronchoalveolar Lavage in Patients With Severe SARS-CoV-2 Infection
Brief Title: Incidence of VAP in Patients With Severe COVID-19
Acronym: CoV-AP
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 20/01/2021-0002005-U
Record Dates: First submitted 2021-01-27; First posted 2021-02-23 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Ventilator Associated Pneumonia; Covid19
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab, Bronchial aspirate, bronchoalveolar lavage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- VAP - BAL positive: Clinically suspected VAP, microbiologically confirmed by BAL
  Interventions: Diagnostic Test: bronchoalveolar lavage
- VAP - BAL negative: Clinically suspected VAP, not microbiologically confirmed by BAL
  Interventions: Diagnostic Test: bronchoalveolar lavage
- NO VAP: No clinically suspected VAP during mechanical ventilation

INTERVENTIONS:
Diagnostic Test: bronchoalveolar lavage — BAL and ETA are performed as per clinical practice on clinical suspicion of VAP (Johanson score)
  Groups: VAP - BAL negative; VAP - BAL positive

SUMMARY:
Combined retrospective and prospective cohort study to evaluate the incidence of microbiologically confirmed VAP in mechanically ventilated patients with COVID-19. In the retrospective part, microbiological data are based on bi-weekly surveillance ETA. In the prospective part, microbiological data are based on ETA and BAL performed on VAP suspicion. In the prospective part, immunological and virological analyses will be performed on biological samples (blood, respiratory tract) collected from patients at VAP diagnosis.

DETAILED DESCRIPTION:
Ventilator-associated pneumoniae (VAP) is the most common infection acquired in the intensive care unit (ICU). To date, there is no diagnostic gold standard for VAP, and its diagnosis is based on scores that include radiologic, clinical, laboratory, and microbiologic parameters. In addition, there is no univocal recommendation regarding the type of microbiological diagnostics. Some guidelines suggest the use of noninvasive methods (endotracheal aspiration, ETA) with semiquantitative cultures, while others suggest the collection of distal respiratory samples (bronchoalveolar lavage, BAL) with quantitative cultures. While the former method is characterized by higher sensitivity and lower specificity, the latter in contrast has higher specificity. To date, there is no evidence that one method is superior to the other in terms of clinical outcome.

In patients with severe SARS-CoV-2 infection, COVID-19 disease itself and immunomodulatory therapies have a direct impact on most of the clinical, laboratory and radiologic parameters required to achieve VAP diagnosis. In this setting, a diagnostic approach characterized by higher sensitivity coupled with lower specificity could lead to of a high number of false positives. The greatest risk is that of an overdiagnosis of VAP and a consequent overtreatment, with the related therapeutic toxicity and increased antibiotic resistance.

At the investigators' Hospital, the diagnosis of VAP is based on clinical-radiological suspicion according to the Johanson score (new finding or progression of infiltrates on lung radiography + at least two of the following three clinical criteria: fever > 38°C, leukocytosis or leukopenia, purulent secretions), widely validated in non-COVID patients. Until the end of 2020, microbiological data to confirm the diagnosis of clinically suspected VAP and to guide antibiotic therapy were based on the performance of biweekly surveillance ETA. In view of the limited specificity of this approach in COVID-19 setting, from the end of 2020 patients with SARS-CoV-2 infection and suspected VAP undergo, if clinically possible, to collection of distal respiratory specimens by performing BAL/mini-BAL.

The present prospective-retrospective cohort study aims to evaluate the incidence of microbiologically confirmed VAP with BAL (prospective part) and biweekly surveillance ETA (retrospective part) in mechanically ventilated patients with COVID-19 in the ICU. In the prospective part, immunological and virological analyses will be performed on biological samples (blood, respiratory tract) collected from patients at VAP diagnosis.

The study will last 12 months.

ELIGIBILITY:
Retrospective part all patients admitted to the ICU for COVID-19-related respiratory failure since the beginning of the pandemics will be included.

Prospective part

Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of SARS-CoV-2 infection by means of reverse transcription polymerase chain reaction (RT-PCR)
* Respiratory failure requiring mechanical ventilation
* mechanical ventilation ongoing for less than 48h

Exclusion Criteria:

* Age < 18 years
* mechanical ventilation ongoing for more than 48h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients with severe SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of VAP | 1,000 ventilator days
  Incidence of clinically suspected and microbiologically confirmed VAP by means of BAL

SECONDARY OUTCOMES:
number of episodes with concordance in bacterial isolates between BAL and ETA performed on VAP suspicion | 1,000 ventilator days
  microbiological concordance of respiratory specimens collected by BAL and ETA on VAP suspicion
number of episodes with concordance in bacterial isolates between BAL performed on VAP suspicion and the preceding surveillance ETA | 1,000 ventilator days
  microbiological concordance of respiratory specimens collected by BAL on VAP suspicion and the preceding bi-weekly surveillance ETA
number of episodes with concordance in cellular phenotype between BAL and peripheral blood on VAP suspicion | 1,000 ventilator days
  immunological analysis of cellular phenotype in BAL and peripheral blood collected on VAP suspicion
number of episodes with concordance in lymphocyte-monocyte activation between BAL and peripheral blood on VAP suspicion | 1,000 ventilator days
  immunological analysis of lymphocyte-monocyte activation in BAL and peripheral blood collected on VAP suspicion
number of episodes with concordance in SARS-CoV-2 viral quantification between BAL, ETA and nasopharyngeal swab on VAP suspicion | 1,000 ventilator days
  virological analysis of SARS-CoV-2 viral quantification in BAL, ETA and nasopharyngeal swab collected on VAP suspicion (subgroup analysis)
number of episodes with concordance in SARS-CoV-2 sequencing between BAL, ETA and nasopharyngeal swab on VAP suspicion | 1,000 ventilator days
  virological analysis of SARS-CoV-2 sequencing in BAL, ETA and nasopharyngeal swab collected on VAP suspicion (subgroup analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Grasselli, MD, Principal Investigator — Intensive Care Unit, IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation; Andrea Gori, MD, Principal Investigator — Infectious Diseases Unit, IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation; Mauro Panigada, MD, Principal Investigator — Intensive Care Unit, IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation; Alessandra Bandera, MD, PhD, Principal Investigator — Infectious Diseases Unit, IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation
Locations (1):
- IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be shared upon written request to the study director

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Background] Rosenthal VD, Al-Abdely HM, El-Kholy AA, AlKhawaja SAA, Leblebicioglu H, Mehta Y, Rai V, Hung NV, Kanj SS, Salama MF, Salgado-Yepez E, Elahi N, Morfin Otero R, Apisarnthanarak A, De Carvalho BM, Ider BE, Fisher D, Buenaflor MCSG, Petrov MM, Quesada-Mora AM, Zand F, Gurskis V, Anguseva T, Ikram A, Aguilar de Moros D, Duszynska W, Mejia N, Horhat FG, Belskiy V, Mioljevic V, Di Silvestre G, Furova K, Ramos-Ortiz GY, Gamar Elanbya MO, Satari HI, Gupta U, Dendane T, Raka L, Guanche-Garcell H, Hu B, Padgett D, Jayatilleke K, Ben Jaballah N, Apostolopoulou E, Prudencio Leon WE, Sepulveda-Chavez A, Telechea HM, Trotter A, Alvarez-Moreno C, Kushner-Davalos L; Remaining authors. International Nosocomial Infection Control Consortium report, data summary of 50 countries for 2010-2015: Device-associated module. Am J Infect Control. 2016 Dec 1;44(12):1495-1504. doi: 10.1016/j.ajic.2016.08.007. Epub 2016 Oct 11. PMID 27742143
- [Background] Papazian L, Klompas M, Luyt CE. Ventilator-associated pneumonia in adults: a narrative review. Intensive Care Med. 2020 May;46(5):888-906. doi: 10.1007/s00134-020-05980-0. Epub 2020 Mar 10. PMID 32157357
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Executive Summary: Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):575-82. doi: 10.1093/cid/ciw504. PMID 27521441
- [Background] Torres A, Niederman MS, Chastre J, Ewig S, Fernandez-Vandellos P, Hanberger H, Kollef M, Li Bassi G, Luna CM, Martin-Loeches I, Paiva JA, Read RC, Rigau D, Timsit JF, Welte T, Wunderink R. International ERS/ESICM/ESCMID/ALAT guidelines for the management of hospital-acquired pneumonia and ventilator-associated pneumonia: Guidelines for the management of hospital-acquired pneumonia (HAP)/ventilator-associated pneumonia (VAP) of the European Respiratory Society (ERS), European Society of Intensive Care Medicine (ESICM), European Society of Clinical Microbiology and Infectious Diseases (ESCMID) and Asociacion Latinoamericana del Torax (ALAT). Eur Respir J. 2017 Sep 10;50(3):1700582. doi: 10.1183/13993003.00582-2017. Print 2017 Sep. PMID 28890434
- [Derived] Mangioni D, Panigada M, Palomba E, Bobbio C, Chatenoud L, Alagna L, Fumagalli J, Gori A, Grancini A, Guzzardella A, Lombardi A, Matinato C, Meli A, Muscatello A, Porretti L, Tomasello M, Trombetta E, Valenti L, Bandera A, Grasselli G. Incidence, microbiological and immunological characteristics of ventilator-associated pneumonia assessed by bronchoalveolar lavage and endotracheal aspirate in a prospective cohort of COVID-19 patients: CoV-AP study. Crit Care. 2023 Sep 26;27(1):369. doi: 10.1186/s13054-023-04658-5. PMID 37749631
- See also: COVID-19 cases worldwide — http://systems.jhu.edu